CLINICAL TRIAL: NCT05506397
Title: The Effect of Acupressure on Constıpatıon Symptoms and Quality of Lıfe in Elderly People
Brief Title: Acupressure for Constipation in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Nigde Omer Halisdemir University (Other); Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba AYDEMİR, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ErciyesU2
Record Dates: First submitted 2022-07-23; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Constıpatıon
Keywords: Acupressure; Constipation; Quality of life; Elderly people; Nursing
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, pretest-posttest control group study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A double-blind design was applied, including participants, interviewers and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (intervention group) (Experimental): Acupressure was applied to individuals in the acupressure group every day for 12 days.
  Interventions: Other: Acupressure
- control group (Placebo Comparator): Placebo acupressure was applied to the individuals in the placebo acupressure group in accordance with the same protocol.
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — Acupressure is a technique based on stimulating certain points on the body with stimulation methods such as hands and fingers.

SUMMARY:
This study was carried out to determine the effect of acupressure applied to LI4, CV12, ST25 and ST36 acupuncture points for a total of 21 minutes, three to each point, on the symptoms of constipation and quality of life of elderly individuals.

DETAILED DESCRIPTION:
The study is a qualitative and quantitative mixed method, double-blind, randomized, placebo-controlled, pretest-posttest control group study. In this study; a total of 81 elderly individuals over the age of 65 and diagnosed with constipation in a family health center were included, 41 individuals in the acupressure group and 40 individuals in the placebo control group. Ethics committee approval, informed voluntary consent of the elderly and all other necessary permissions to conduct the study were obtained before the study.

The data of the study were collected using the Individual Identification Form, the Constipation Assessment Scale (CAS), the Constipation Quality of Life Scale (PAC-QOL), the Visual Analog Scale (VAS), the Individual Follow-up Form and the Semi-Structured Interview Form. Acupressure was applied to individuals in the acupressure group every day for 12 days, and placebo acupressure was applied to individuals in the placebo acupressure group at the same time and in line with the same protocol. In addition, individual in-depth interviews were conducted with the individuals in the acupressure group after the applications were completed.

Quantitative data were evaluated using the IBM SPSS Statistics for Windows 24.0 package program. In the evaluation of quantitative data; Independent groups t test / Mann Whitney U test, dependent groups t-test, two-way mixed pattern ANOVA, multiple regression analysis (enter method) were used and p<0.05 value was considered statistically significant. In the evaluation of qualitative data, descriptive and content analysis methods were used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and over,
* Able to answer cognitive questions
* Able to do daily tasks unaided
* Experiencing two or more of the Rome IV criteria

Exclusion Criteria:

* Communication and adaptation difficulties,
* Malignant, intestinal obstruction, fecal incontinence, diarrhea, irritable bowel syndrome, abdominal infection, etc. have a contraindication to continue the intervention, addicted to bed
* Chronic pain requiring long-term analgesic intake and using psychiatric medication,

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Constipation Assessment Scale (CAS) | Change from Baseline symptoms of constipation at 12 days
  It was used to evaluate the symptoms of constipation.

SECONDARY OUTCOMES:
Constipation Quality of Life Scale (PAC-QOL) | Change from baseline constipation-related quality of life at 12 days
  It was used to evaluate the quality of life.
Visual Analog Scale (VAS) | Change from baseline defecation comfort at 12 days
  It was used to assess the level of defecation comfort.
Number of Defecation | Change from baseline number of defecations at 12 days
  12-day total number of defecations

CONTACTS AND LOCATIONS:
Overall Officials: Sultan TAŞCI, Prof. Dr., Study Director — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Kayseri̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: unlimited
Access Criteria: unlimited

REFERENCES:
- [Background] Shin J, Park H. Effects of Auricular Acupressure on Constipation in Patients With Breast Cancer Receiving Chemotherapy: A Randomized Control Trial. West J Nurs Res. 2018 Jan;40(1):67-83. doi: 10.1177/0193945916680362. Epub 2016 Nov 30. PMID 27903827
- [Background] Wang PM, Hsu CW, Liu CT, Lai TY, Tzeng FL, Huang CF. Effect of acupressure on constipation in patients with advanced cancer. Support Care Cancer. 2019 Sep;27(9):3473-3478. doi: 10.1007/s00520-019-4655-1. Epub 2019 Jan 24. PMID 30675666
- [Background] Jung ES, Chang AK. Effects of Auricular Acupressure in Patients on Hemodialysis. J Nurs Res. 2020 Aug;28(4):e106. doi: 10.1097/jnr.0000000000000378. PMID 32379107
- [Result] Lee EJ, Frazier SK. The efficacy of acupressure for symptom management: a systematic review. J Pain Symptom Manage. 2011 Oct;42(4):589-603. doi: 10.1016/j.jpainsymman.2011.01.007. Epub 2011 Apr 30. PMID 21531533
- [Derived] Aydemir T, Tasci S, Bayraktar M, Saz A. The effect of acupressure on constipation symptoms and quality of life among older people: a mixed-methods study. Eur Geriatr Med. 2023 Oct;14(5):1135-1144. doi: 10.1007/s41999-023-00842-6. Epub 2023 Jul 21. PMID 37477804
- Available data/document: Clinical Study Report — https://tez.yok.gov.tr/UlusalTezMerkezi/